CLINICAL TRIAL: NCT03739151
Title: Applying Novel Passive Sensing Technology to Target Adherence to Diet in Behavioral Obesity Treatment for Patients With Cardiovascular Disease Risk
Brief Title: Passive Sensing Technology for Lapse Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Graham Thomas, Associate Professor (Research), The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1F32HL143954-01 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Overweight and Obesity
Keywords: overweight and obesity; eating behavior; nonadherence, patient; ecological momentary assessment; passive sensing; dietary assessment
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Patient Compliance

STUDY DESIGN:
Intervention Model Description: All participants in this study receive gold-standard behavioral obesity treatment on an individual basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Obesity Treatment (Other): All participants will receive gold-standard behavioral obesity treatment
  Interventions: Behavioral: Behavioral Obesity Treatment

INTERVENTIONS:
Behavioral: Behavioral Obesity Treatment — Self-monitoring. Participants will be taught to record their weight, the calories of each food item, and physical activity using a method of their choice (e.g., commercial smartphone app, paper diary). The clinician will review dietary intake and provide personalized feedback at the outset of session.
  Diet. Per national guidelines for weight loss, a daily goal of 1200-1800 kcal/day will be prescribed depending on baseline weight. A Mediterranean diet will be prescribed to meet the recommended calorie goal and be consistent with dietary recommendations for CVD patients.
  Exercise. Participants will be encouraged to achieve 250 minutes/week of moderate intensity activity in accordance with current national recommendations for physical activity among individuals attempting weight loss. Participants will be encouraged to gradually increase activity level to achieve approximately 50 minutes of activity over five days per week.
  Other Names: Behavioral Weight Loss

SUMMARY:
Behavioral obesity treatment (BOT) produces clinically significant weight loss and health benefits for many individuals with overweight/obesity and cardiovascular disease (CVD). Yet, about half of patients fall short of expected outcomes and most experience gradual weight regain, thus negating the benefits over time. Lapses (i.e., self-reported eating instances that deviate from the BOT prescribed diet) could explain poor outcomes, but the behavior is understudied because it is difficult to assess in-lab and via self-report. The investigators therefore propose to study lapses using a multimethod approach with the following tools: ecological momentary assessment (EMA; repeated sampling method via mobile device), a wrist-worn device that automatically detects eating behavior and various eating characteristics (frequency, rate, and duration of eating episodes), and 24-hour dietary recalls. The investigators will recruit participants (n=40) with overweight/obesity and one additional CVD risk factor to enroll in a 12-week BOT program and an additional 12-week period of weight loss maintenance. Participants will complete a biweekly 7-day EMA protocol to self-report on eating behavior, including the occurrence of dietary lapse. Participants will continuously wear the wrist-worn ActiGraph Link to characterize eating behavior. Lastly, participants will complete 24-hour dietary recalls via structured interview (split between days with and without lapses) at 6-week intervals to measure the composition of all food and beverages consumed. This study aims to 1) identifying characteristics of lapse behavior by measuring passively-sensed timing, duration, frequency, and rate of eating amongst known lapse episodes, 2) test the association between dietary lapse frequency and weight change, and 3) estimate nutrition composition of dietary lapses. The study approach is consistent with priorities of NHLBI to optimize clinical research and diagnostic strategies to improve CVD and related risk factors.

DETAILED DESCRIPTION:
Design and overview. This proposal adds continuous passive sensing and periodic dietary assessment to EMA to measure dietary lapses in adults with overweight/obesity and CVD risk (n=40) throughout a BOT program (12 weeks) and a period of weight loss maintenance (12 weeks). Participants will self-report via EMA on meals and snacks, indicting when dietary lapses occur. The ActiGraph Link, a wrist-worn device that can detect the motion of food being brought to the mouth, will be used to objectively detect eating characteristics. Because the composition of foods consumed during lapses is an important facet of lapse behavior that is not measured well via passive sensing or EMA, participants will complete periodic 24-hour dietary recalls via structured interview (split between days with and without lapses) to measure the composition of all food and beverages consumed. Data from the EMA, ActiGraph, and food recalls will be integrated to assess characteristics (i.e., frequency, rate, duration), estimated caloric content, and composition of dietary lapses compared to non-lapses. The study will advance the science of weight control by combining gold-standard and innovative methods to objectively measure dietary lapses and test their association with weight change in BOT.

Recruitment and Screening. Participants will be recruited on a rolling basis using advertisements in local newspapers, the study Center's website, and advertising resources available through the Miriam Hospital. The study will recruit over 12 months aiming for 4 participants per month. Interested individuals will be contacted via telephone to complete initial screening. The study procedures will be summarized, and an in-person appointment will be scheduled for additional screening and orientation. At the orientation meeting, a thorough overview of the study purpose and procedures will be provided and consent obtained. Consented individuals will be asked to complete all screening questions and measures to determine eligibility. Eligible participants will be contacted after this visit to begin treatment. Ineligible individuals will be notified accordingly and provided with referrals for BOT in the community.

The behavioral obesity treatment is described in further detail below.

Assessment schedule. Measures are described in further detail below. The primary outcome of interest, dietary lapse, will be measured on a biweekly basis throughout the 24-week study. Participants will continuously wear a wrist-watch device to passively detect eating episodes. Composition and quality of dietary intake will be measured every 6 weeks. Participants will have weight measured and wrist-watch data downloaded at each weekly appointment during the weight loss treatment phase. During the maintenance phase of treatment, participants will be asked to attend an additional appointment once per month separate from the monthly treatment visit, to initiate data downloading on the wrist-watch sensor and have weight measured.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (body mass index 25-45 kg/m2)
* Interested and able to participate in in-person weight loss intervention
* Physician-diagnosed one or more CVD risk factors (type 2 diabetes/prediabetes, hypercholesterolemia, or hypertension).

Exclusion Criteria:

* Report health problems that preclude weight loss or physical activity
* Are currently pregnant or breastfeeding, or planning to be pregnant within the next 6 months,
* Are currently or recently (< 6 months) enrolled in a commercial weight loss program
* Have lost ≥ 5% of their initial body weight in the last 6 months
* Currently taking weight loss medication
* Have had a previous surgical procedure for weight loss
* Have a history of a clinically diagnosed eating disorder excluding Binge Eating Disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Sensor-based Dietary Lapse | 24-week frequency of sensor-based dietary lapse
  Participants will wear a wrist-worn 9-axis accelerometer during waking hours that measures wrist-roll motion, which can objectively assess dietary lapses.

SECONDARY OUTCOMES:
Self-reported Dietary Lapse | Participants will be asked to complete 7 days of EMA on a biweekly basis for 24 weeks. Therefore, participants will complete EMA at weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23.
  Lapses will be assessed via ecological momentary assessment (EMA), a repeated sampling method using electronic forms on smartphone devices.
Weight | Weight will be measured at each study appointment (baseline assessment, weekly for 12 weeks, and twice monthly for the subsequent 12 weeks).
  Participants' body weight will be measured to the nearest 0.1 kg using a calibrated digital scale
Dietary Composition | Dietary composition will be assessed at baseline and at weeks 5, 11, 17, and 23
  Dietary composition will be assessed using 24-hour food recall method. The Nutrition Data System for Research (NDSR), a computer-based software application developed at the University of Minnesota Nutrition Coordinating Center (NCC) will facilitate the collection of recalls in a standardized fashion

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thomas, PhD, Study Chair — The Miriam Hospital; Stephanie P Goldstein, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
The raw data from the current project are too large to easily transfer to individual investigators. As such, the investigators plan to develop a cost-effective, safe plan for sharing de-identified participant data upon reasonable request by other researchers.

REFERENCES:
- [Derived] Goldstein SP, Olson KL, Thomas JG. Association of weight and shape concern with weight change and weight-related behaviors in behavioral weight loss treatment. J Behav Med. 2023 Dec;46(6):1049-1056. doi: 10.1007/s10865-023-00451-5. Epub 2023 Sep 23. PMID 37740874
- [Derived] Goldstein SP, Hoover A, Thomas JG. Combining passive eating monitoring and ecological momentary assessment to characterize dietary lapses from a lifestyle modification intervention. Appetite. 2022 Aug 1;175:106090. doi: 10.1016/j.appet.2022.106090. Epub 2022 May 20. PMID 35598718
- [Derived] Goldstein SP, Hoover A, Evans EW, Thomas JG. Combining ecological momentary assessment, wrist-based eating detection, and dietary assessment to characterize dietary lapse: A multi-method study protocol. Digit Health. 2021 Feb 2;7:2055207620988212. doi: 10.1177/2055207620988212. eCollection 2021 Jan-Dec. PMID 33598309

DOCUMENTS (1):
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03739151/ICF_000.pdf